CLINICAL TRIAL: NCT03578003
Title: Morning Bright Light to Improve Sleep Quality in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Miranda M Lim, Staff Physician and Assistant Professor, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4085
Record Dates: First submitted 2018-06-13; First posted 2018-07-05 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Brain Injuries, Traumatic; Post-traumatic Stress Disorder
Keywords: Sleep; Bright Light
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Bright Light Therapy (Experimental): Subjects who engage in morning bight light therapy
  Interventions: Other: Morning Bright Light Therapy
- Control (No Intervention): Subjects who do not engage in morning bright light therapy

INTERVENTIONS:
Other: Morning Bright Light Therapy — 60 minutes of bright light therapy (10,000 lux) received within 90 minutes of waking
  Arms: Morning Bright Light Therapy

SUMMARY:
One of the principal complicating factors associated with traumatic brain injury (TBI) is sleep-wake disturbances (e.g., insomnia, excessive daytime sleepiness, and circadian rhythm sleep disorders). Morning bright light therapy (MBLT) has been shown to improve sleep quality in a variety of conditions, but little has been done investigating the utility of MBLT in improving sleep in Veterans with TBI. This proposal aims to determine the effect of MBLT on sleep quality in Veterans with TBI. Veterans with and without TBI will be recruited from the VA Portland Health Care System. Baseline questionnaires and 7 days of actigraphy will be collected prior to engaging in 60 minutes of MBLT daily for 4 weeks, during which actigraphy will also be collected continuously. Post-MBLT questionnaire data will be collected, and follow-up questionnaire data will be collected at 3 months post-MBLT.

ELIGIBILITY:
Inclusion Criteria:

* Veterans

Exclusion Criteria:

* History of bipolar disorder
* History of macular degeneration
* Non-English speaking
* Decisionally impaired
* Currently using a light box

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline; after 4 weeks of intervention; and 2 months after the end of intervention
  Measures self-reported insomnia severity; total score range = 0-28 (higher total score = worse insomnia)

CONTACTS AND LOCATIONS:
Overall Officials: Miranda M Lim, MD, PhD, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Health Care System, Portand, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifiable data will be made available to qualified researchers on request to the study PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Information will be sent as soon as is practical and will be available as long as the PI is available.
Access Criteria: Legitimate research agenda, including but not limited to request to double-check presented or published results and novel analyses.

REFERENCES:
- [Derived] Elliott JE, McBride AA, Balba NM, Thomas SV, Pattinson CL, Morasco BJ, Wilkerson A, Gill JM, Lim MM. Feasibility and preliminary efficacy for morning bright light therapy to improve sleep and plasma biomarkers in US Veterans with TBI. A prospective, open-label, single-arm trial. PLoS One. 2022 Apr 14;17(4):e0262955. doi: 10.1371/journal.pone.0262955. eCollection 2022. PMID 35421086